CLINICAL TRIAL: NCT05538221
Title: Reliability of a Low-cost Video-based Gait Analysis System
Brief Title: Reliability of a Gait Analysis System
Status: Completed | Type: Observational
Sponsor: Centro Integral de Neurologia y Especialidades Afines, Argentina (Other)
Collaborators: Fundación Favaloro (Unknown); Institut Guttmann (Other)
Responsible Party: Principal Investigator, Bernardo Centeno, Medical Doctor, Centro Integral de Neurologia y Especialidades Afines, Argentina
Other Study IDs: ConfSilema; NCT05305755 (obsolete NCT alias)
Record Dates: First submitted 2022-09-09; First posted 2022-09-13 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Gait Analysis
Keywords: Gait; Reliability; Video; Kinematics; Temporo Spatial Parameters

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: SILEMA — SILEMA consists of a webcam connected to a laptop, a LED reflector, and a software. To carry out gait analysis with SILEMA, an Evaluator must place six yellow auto-adhesive markers over certain anatomical landmarks in the lower limbs, namely, greater trochanter, external femoral condyle, head of the fibula, lateral malleolus and base and head of the fifth metatarsal. The patient is asked to walk barefoot through an eight meter walkway at a self-selected speed, while a webcam connected to a laptop records a video. Then, an Operator, making use of the software, processes the video, obtaining spatio-temporal and joint kinematic parameters.

SUMMARY:
Gait disturbances can be observed in all age groups, and may be due to different conditions, such as advanced age, stroke, head trauma, spinal cord injury, cerebral palsy, myelomeningocele, among others. The aforementioned gait disorders are associated with an increased risk of falls (which can cause major fractures or head trauma), decreased mobility, loss of independence, cardiovascular pathology, and decreased quality of life. In order to improve a given abnormal gait pattern, an objective assessment of gait is necessary. There are several methods to carry out gait evaluations, like Instrumented Gait Analysis (High cost, time-consuming, qualified professionals needed) and the ones based on observation (limited reliability and validity). An alternative, is the use of video-based systems. SILEMA (Computer System for Gait Study Laboratories in Argentina) is a video-based low-cost gait analysis system that measures temporo-spatial (speed, step length, cadence, stance and swing times) and joint kinematic (Hip, Knee, Ankle) parameters. Its reliability has not been reported yet; thus the primary aim of this study is to determine both the "intra-evaluator" (same evaluator, different sessions) and "inter-evaluator" (same session, different evaluators) reliability.

DETAILED DESCRIPTION:
Gait disturbances can be observed in all age groups, and may be due to different conditions, such as advanced age, stroke, head trauma, spinal cord injury, cerebral palsy, myelomeningocele, among others. The aforementioned gait disorders are associated with an increased risk of falls (which can cause major fractures or head trauma), decreased mobility, loss of independence, cardiovascular pathology, and decreased quality of life.

One of the main objectives of rehabilitation is the improvement of the gait pattern, for which a correct evaluation of it is a necessary condition. Gait analysis is the systematic study of human locomotion, with joint kinematics (description of movement in different planes) and temporo-spatial parameters (speed, cadence, step length, stance and swing times) being variables usually valued and reported. There are several methods for conducting gait assessments. One of them consists of the administration of scales based on observation, which are accessible and simple to execute, but exhibit limited reliability and validity, depending in addition to the previous experience of the observer. The method considered "Gold standard" is the Instrumented Gait Analysis (IGA), from which parameters of kinematics (through optoelectronic cameras and reflective markers), kinetics (through the use of force platforms) and muscle activity (using electromyography) can be obtained.Unfortunately, these systems are not available in most rehabilitation centers, due to the high cost they represent, the need to have highly trained professionals for their use and the long time needed for calibration and post-processing, difficulties that are continuously mentioned in the literature. An alternative to IGA is the use of video-based systems that allow the quantification of temporo-spatial parameters and joint kinematics. One of these systems is SILEMA(Computer System for Gait Study Laboratories in Argentina) which is based on the technique of digital videography. This system exhibits the advantages of being portable, easy to implement and use, and low cost.The purpose of the clinical analysis of gait is usually to differentiate between normal and abnormal patterns, and to assess the change over time or due to an intervention (surgery, orthosis, botulinum toxin, physical therapy, etc.), being necessary in the latter case to make repeated measurements. Usually, to carry out gait evaluations, the patient is asked to perform several "passes", each of them consisting of a free gait through a walkway, at a "self-selected" speed, during a session in which the corresponding information is collected. In healthy subjects, there is usually a variability between repeated measurements (both intra-subject and inter-subject), which occurs at the expense of intrinsic factors (age, height, gait speed, etc.) or extrinsic, caused by methodological errors (experimental error), such as those related to the placement of markers (task carried out by an evaluator, usually a Therapist, or with the processing of a video made by the operator of the software. The consistency or repeatability of the measurements is what is known as reliability. In other words, reliability is a measure of the variability that exists between repeated measurements, and is usually estimated, as recommended, using the intraclass correlation coefficient "ICC" (Relative Reliability) and the standard error of the measure "SEM" (Absolute Reliability). Its determination is very important, since in daily practice it could give information on whether the observed change in a certain parameter of the gait is due to the intervention / evolution of the pathology or to the variability of the measurements. In the context of gait analysis, reliability is typically evaluated "inter-pass" (between several passes of the same subject, in the same session), "intra-operator" (same video evaluated by the same operator at two different times), "interoperator" (same video, different operators), "intra-evaluator" (same evaluator, different sessions) and "inter-evaluator" (same session, different evaluators). To the best of our knowledge, the reliability of SILEMA has not been reported, being the objective of the present study, to determine this metric, with the intention of expanding its use, both for the clinic and for research.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years

Exclusion Criteria:

* History of any condition (neuromuscular, cardiovascular and/or musculoskeletal) that could generate an atypical gait pattern
* Pregnancy
* Known hypersensitivity to adhesive tape

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adult volunteers
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2022-11-04 (Actual); Study Completion 2022-11-04 (Actual)

PRIMARY OUTCOMES:
Step Length | One Week
  Distance between the initial contact of one foot, and the next initial contact of the other foot, expressed in meters. Kinematic parameter to define reliability
Speed | One Week
  Distance travelled in the unit of time, expressed in meters/seconds .Kinematic parameter to define reliability
Cadence | One Week
  Number of steps performed on the unit of time. Kinematic parameter to define reliability
Stance Time | One Week
  Time elapsed between the initial contact of one foot and the take-off of the toes of the same foot, expressed in seconds.Kinematic parameter to define reliability
Swing Time | One Week
  Time elapsed between take-off of the toes and the next initial contact of the same foot, expressed in seconds. Kinematic parameter to define reliability
Hip Range of Motion | One Week
  In Degrees. Kinematic parameter to define reliability
Knee Range of Motion | One Week
  In Degrees. Kinematic parameter to define reliability
Ankle Range of Motion | One Week
  In Degrees. Kinematic parameter to define reliability
Minimum Hip angle | One Week
  In Degrees. Kinematic parameter to define reliability
Minimum Knee angle | One Week
  In Degrees. Kinematic parameter to define reliability
Minimum Ankle angle | One Week
  In Degrees. Kinematic parameter to define reliability
Maximum Hip angle | One Week
  In Degrees. Kinematic parameter to define reliability
Maximum Knee angle | One Week
  In Degrees. Kinematic parameter to define reliability
Maximum Ankle angle | One Week
  In Degrees. Kinematic parameter to define reliability

CONTACTS AND LOCATIONS:
Overall Officials: Bernardo Centeno, Principal Investigator — Centro Integral de Neurologia y Especialidades Afines, Argentina
Locations (1):
- CINEA, San Miguel de Tucumán, Tucumám, Argentina

IPD SHARING:
Plan to Share IPD: Undecided